CLINICAL TRIAL: NCT01777451
Title: Whole Body Magnetic Resonance Imaging With Diffusion Weighted Imaging : Potential Role in Neurofibromatosis
Acronym: NEFIMAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Steven Pans, Medical Doctor Radiologist, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: NEFIMAR; S52684 (Other: Clinicla trial Center UZ Leuven)
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Whole Body Imaging; Magnetic Resonance Imaging; Neurofibromatosis 1; Diffusion Magnetic Resonance Imaging; Peripheral Nerve Sheath Tumors, Malignant
Keywords: Whole Body Imaging; Magnetic Resonance Imaging; Neurofibromatosis 1; Diffusion Magnetic Resonance Imaging; Peripheral Nerve Sheath Tumors, Malignant
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibrosarcoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neurofibromatosis 1: All patients diagnosed with neurofibromatosis type 1. GROUP 1:ADDITIONAL IMAGING OR SURGERY There will be patients with high-risk neurofibromas (potential malignant). These patients will underwent additional examinations or surgery (outside this study). Follow-up MRI within 2 years (study MRI )
  GROUP 2:
  No suspicious lesions at MRI. Follow-up within 2 years(Study MRI).
  Interventions: Other: Additional imaging or surgery

INTERVENTIONS:
Other: Additional imaging or surgery — No specific intervention is necessary. If a suspicious lesion is diagnosed on MRI, further investigation will be planned (PET-CT or surgery - biopsy)

SUMMARY:
Whole body MRI will be performed in patients with neurofibromatosis Type 1

PURPOSE 1:

To determine the total tumor load (neurofibroma) and to diagnose plexiform neurofibromas or malignant peripheral nerve sheath tumors. All patients will be scanned two years after the baseline whole body MRI to investigate to investigate the changes of total tumor load.

PURPOSE 2: added value of diffusion weighted imaging in diagnosis of high-risk neurofibromas

PURPOSE 3 : to determine the apparent diffusion coefficient of the malignant nerve sheath tumors and neurofibroma.

PURPOSE 4 : correlation between histopathology of the surgically resected neurofibroma/malignant nerve sheath tumors and MRI findings

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurofibromatosis type 1, between 6 and 50 years old

Exclusion Criteria:

* Patients who are not allowed to be scanned on MRI (contra-indications: pacemaker ed.)

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients with a clinically proven neurofibromatosis type 1 can be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Estimation of total tumor load and diagnosis of high-risk neurofibromas | 1 month
  Estimation of the total tumor load of neurofibromas with whole body MRI (head to knee). Diagnosis of high risk neurofibroma in the chest, abdomen, pelvis, and extremities with T2-weighted sequence and diffusion weighted sequence.

SECONDARY OUTCOMES:
To diagnose high-risk neurofibroma | 2 months
  Some patients with neurofibromatosis have lesions, pre-malignant or malignant neurofibromas. Additional imaging (PET-CT), a biopsy or surgical treatment is necessary in combination with histopathology of the lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pans, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Tucker T, Friedman JM, Friedrich RE, Wenzel R, Funsterer C, Mautner VF. Longitudinal study of neurofibromatosis 1 associated plexiform neurofibromas. J Med Genet. 2009 Feb;46(2):81-5. doi: 10.1136/jmg.2008.061051. Epub 2008 Oct 17. PMID 18930997
- [Background] Cai W, Kassarjian A, Bredella MA, Harris GJ, Yoshida H, Mautner VF, Wenzel R, Plotkin SR. Tumor burden in patients with neurofibromatosis types 1 and 2 and schwannomatosis: determination on whole-body MR images. Radiology. 2009 Mar;250(3):665-73. doi: 10.1148/radiol.2503080700. PMID 19244040
- [Background] Van Meerbeeck SF, Verstraete KL, Janssens S, Mortier G. Whole body MR imaging in neurofibromatosis type 1. Eur J Radiol. 2009 Feb;69(2):236-42. doi: 10.1016/j.ejrad.2008.10.024. Epub 2008 Dec 16. PMID 19091504